CLINICAL TRIAL: NCT01841476
Title: POL6326 - A Phase I, Open, Single Intravenous Infusion Dose, Pharmacokinetic and Pharmacodynamic Study in Healthy Volunteers Who Are Volunteering as Haematopoietic Stem Cell (HSC) Donors
Brief Title: Safety and Efficacy of POL6326 for Mobilization of Hematopoietic Stem Cells in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Polyphor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POL-3
Record Dates: First submitted 2013-04-02; First posted 2013-04-26 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Peripheral blood; HSC; Mobilization; CXCR4; volunteers
MeSH Terms: interventions — balixafortide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- POL6326 (Experimental): 2-hour single intravenous infusion doses of POL6326
  Interventions: Drug: POL6326

INTERVENTIONS:
Drug: POL6326

SUMMARY:
Phase I study to determine and compare the safety/tolerability of single ascending doses of POL6326 by intravenous infusion.

DETAILED DESCRIPTION:
Phase I Study

* to determine and compare the safety of single ascending doses of POL6326 by intravenous infusion
* to determine the relationship between 2-hour single intravenous infusion doses of POL6326 and the concentration of HSC and mature WBC in peripheral blood using immunophenotypic assays.

ELIGIBILITY:
Inclusion Criteria:

1. Mobilization and collection of hematopoietic stem cells (HSCs) using G-CSF at least 6 weeks but less than 6 months prior to protocol enrollment.
2. Ages greater than or equal to 18 years and less than or equal to 55 years.
3. Normal liver and renal function, normal CBC, normal ECG, normal blood pressure including adequately medically controlled idiopathic arterial hypertension, no other contraindications to mobilized peripheral blood stem cell donation according to WMDA criteria and relevant SOPs at the study site defining additional exclusion criteria for stem cell donation.
4. Subject must be eligible for normal blood donation according to requirements for IDMs as laid out by national law for blood donors.
5. Ability to comprehend the investigational nature of the study and provide informed consent.

Exclusion Criteria:

1. Active infection or history of recurrent infection- hepatitis B and C (HBsAg, Anti-HBc, Anti-HCV), HIV and HTLV-1.
2. History of autoimmune disease such as rheumatoid arthritis, systemic lupus erythematous.
3. History of cancer within the past 5 years excluding basal cell or squamous cell carcinoma of the skin.
4. History of any hematologic disorders including thromboembolic disease.
5. History of cardiac disease such as uncontrolled hypertension, peripheral vascular disease, myocardial infarction, cardiac arrhythmias OR related symptoms such as tachycardia, chest pain, shortness of breath which have required medical intervention OR treatment or a Framingham coronary disease risk prediction score of greater than 10% 10 year coronary heart disease (CHD) risk.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-02; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety of single ascending doses of POL6326 by intravenous infusion according to standard criteria | 2 days
  Safety as measured by the incidence, type and severity of adverse events.

SECONDARY OUTCOMES:
Pharmacokinetic outcome | 24h
  Determine the pharmacokinetic profile of POL6326 following single intravenous administration, e.g. Cmax, AUC, terminal half life and clearance
Mobilisation of CD34+ cells | 2 days
  Time dependent measurement of CD34+ cells during and after infusion of POL6326 in all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Halvard Boenig, M.D. Ph.D, Principal Investigator — German Red Cross Blood Service and Institute for Transfusion Medicine and Immunohematology of the Goethe University, Frankfurt, Germany
Locations (1):
- German Red Cross Blood Service and Institute for Transfusion Medicine and Immunohematology of the Goethe University, Frankfurt, Germany

REFERENCES:
- [Derived] Karpova D, Brauninger S, Wiercinska E, Kramer A, Stock B, Graff J, Martin H, Wach A, Escot C, Douglas G, Romagnoli B, Chevalier E, Dembowski K, Hooftman L, Bonig H. Mobilization of hematopoietic stem cells with the novel CXCR4 antagonist POL6326 (balixafortide) in healthy volunteers-results of a dose escalation trial. J Transl Med. 2017 Jan 3;15(1):2. doi: 10.1186/s12967-016-1107-2. PMID 28049490